CLINICAL TRIAL: NCT07253623
Title: Perceptual-Motor Performance and Neural Conduction Asymmetries in Elite Basketball Players
Brief Title: Perceptual-Motor Performance in Elite Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Recep Soslu, Associate Professor, Karamanoğlu Mehmetbey University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025/2287
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Perceptual Motor Performance and Neural Conduction Asymmetries in Elite Basketball Players
Keywords: Coincidence anticipation timing, nerve conduction, electromyography, perceptual-motor performance, hand dominance, basketball
MeSH Terms: interventions — potassium channel subfamily K member 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coincidence Anticipation Timing (CAT)Task (Experimental): The intervention involved participants performing the Coincidence Anticipation Timing (CAT) task using a Bassin anticipation timer device. The task required athletes to anticipate the arrival of a target light and press a button when it lit up. This procedure was conducted for both the dominant and non-dominant hands. The speed of the light sequence was set to 7 m/s. Surface Electromyography (sEMG) and nerve conduction measurements were recorded concurrently during the task to assess neuromuscular responses to the high-speed perceptual-motor challenge
  Interventions: Behavioral: Coincidence Anticipation Timing (CAT) Task

INTERVENTIONS:
Behavioral: Coincidence Anticipation Timing (CAT) Task — The intervention involved participants performing the Coincidence Anticipation Timing (CAT) task using a Bassin anticipation timer device. The task required athletes to anticipate the arrival of the final target light and press a button when it lit up. This procedure was carried out separately for both the dominant and non-dominant hands. The speed of the light sequence was set to 7 m/s. Surface Electromyography (sEMG) and nerve conduction measurements were recorded concurrently during the task to assess neuromuscular responses to the high-speed perceptual-motor challenge.
  Other Names: Coincidence Anticipation Timing Task; CAT task

SUMMARY:
This study investigated upper-extremity asymmetries in perceptual-motor performance and neural conduction among elite female basketball players, utilizing a one-group pretest-posttest design. Fourteen athletes were assessed on Coincidence Anticipation Timing (CAT) performance (Absolute Error, AE; Variable Error, VE), Surface Electromyography (sEMG) parameters (activation latency and amplitude), and Median/Ulnar nerve conduction characteristics. The analysis revealed a significant main effect of Hand Dominance, with the dominant hand exhibiting superior timing accuracy and consistency (lower AE and VE, p < 0.01), which is potentially attributed to enhanced neuromuscular efficiency stemming from sport-specific training adaptations.

Baseline neural assessments indicated enhanced efficiency in the dominant limb, characterized by shorter nerve conduction latency and higher amplitude. However, the dominant limb was also found to be susceptible to greater maximum errors, supporting the presence of a speed-accuracy trade-off in high-velocity perceptual-motor actions. Post-intervention analyses following the CAT task revealed significant, generalized neuromuscular alterations across both limbs, specifically an increase in latency and a decrease in amplitude (p < 0.001), suggesting task-induced acute neuromuscular strain or fatigue.Furthermore, strong correlations were established between nerve conduction latency and error indices (r = 0.72 to 0.87), emphasizing a direct functional link between peripheral neural transmission speed and perceptual-motor precision. In conclusion, elite basketball players exhibit asymmetrical neural adaptations favoring the dominant limb, yet performance variability is intrinsically tied to peripheral neural efficiency. The findings advocate for the integration of bilateral training strategies and electrophysiological monitoring to optimize performance while concurrently mitigating the risk of overuse-related neural compromise.

DETAILED DESCRIPTION:
This study employed a one-group pretest-posttest design to comprehensively investigate the relationship between perceptual-motor performance, muscle activation characteristics, and peripheral nerve conduction velocity in fourteen elite female basketball players (21.6 years, 2.9 years experience). The primary aim was to determine if faster and more consistent neuromuscular responses are associated with improved Coincidence Anticipation Timing (CAT) performance and to identify potential asymmetries between the dominant and non-dominant upper extremities2. Participants underwent baseline testing (pretest) followed by an intervention phase where they performed the CAT task with synchronous recording of surface Electromyography (sEMG) and motor nerve conduction for the Median and Ulnar nerves. CAT performance was quantified using Absolute Error (AE) and Variable Error (VE).

Statistical analysis, utilizing a 2x2 repeated measures ANOVA, revealed significant effects of Hand Dominance on CAT performance. The dominant hand exhibited significantly lower AE and VE (p<0.01) compared to the non-dominant hand, reflecting superior timing accuracy and consistency, likely due to sport-specific motor specialization and enhanced neural efficiency. This was supported by baseline data showing shorter nerve conduction latency and higher amplitude in the dominant limb. However, the dominant hand also demonstrated greater maximum errors, indicating the presence of a speed-accuracy trade-off under high-speed conditions. Furthermore, post-intervention analyses, conducted immediately following the CAT task, demonstrated acute neuromuscular alterations consistent with strain or fatigue. Specifically, both Distal Motor Latency (DML) and Non-Dominant Motor Latency (NDML) showed significant increases from pre- to post-test, and motor and sensory amplitudes (e.g., DMA, NDMA, DUA, NDUA) decreased significantly (p < 0.001), reflecting a slowing of motor nerve conduction and compromised neuromuscular activation capacity.

Secondary analyses using Pearson correlation coefficients highlighted a critical interdependence between neurophysiological and behavioral outcomes. Strong correlations were observed between nerve conduction latency and error indices (r = 0.72 to 0.87), indicating a direct link between the speed of peripheral neural transmission and perceptual-motor precision. Collectively, the findings underscore that while elite basketball players achieve superior performance via asymmetrical neural adaptations favoring the dominant limb, this advantage is sensitive to acute strain. The study concludes that integrating CAT performance metrics with electrophysiological measures provides a novel, evidence-based framework for understanding the neurophysiological underpinnings of perceptual-motor skill. The strong link between neural parameters and error indices emphasizes the need for training and recovery strategies, such as bilateral training and electrophysiological monitoring, to enhance performance efficiency and mitigate the risk of overuse-related neural strain in high-level athletes.

ELIGIBILITY:
Inclusion Criteria:

* To be a female elite basketball athlete, Participants were required to be acquainted with the test methods

Exclusion Criteria:

* To have no neurological symptoms or history, and no previous head injuries, To have no upper extremity injuries or surgeries within the past 6 months.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Absolute Error (AE) and Variable Error (VE) of Coincidence Anticipation Timing (CAT) | Measured at Baseline (Pre-test) and Immediately Post-intervention (Post-test)
  This measure assesses the perceptual-motor accuracy and consistency between the dominant and non-dominant hands.Absolute Error (AE) quantifies the magnitude of the temporal error, irrespective of the response direction (early or late. Variable Error (VE) quantifies the response consistency across trials.The primary hypothesis tested was the asymmetry in timing performance favoring the dominant limb.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiology Laboratory, Faculty of Sports Sciences, Karamanoğlu Mehmetbey University., Karaman, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD), including CAT performance indices (AE and VE) and electrophysiological parameters (nerve conduction latency and amplitude), will be made available upon reasonable request. Data will be shared with qualified researchers only after the publication of the final study results and contingent upon the execution of a formal Data Sharing Agreement (DSA). To protect participant privacy, the data will be anonymized and stripped of any identifying information. Requests for access should be directed to the Corresponding Author (Assoc.Prof. Dr. Recep Soslu) and are subject to approval by the Principal Investigator and the Ethics Committee of Karamanoğlu Mehmetbey University
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date 12/2025 End Date 12/2015
Access Criteria: Access will be granted only to qualified researchers who submit a reasonable research proposal that is consistent with the initial study's objectives or adds significant scientific value. Access is contingent upon the execution of a formal Data Sharing Agreement (DSA) to ensure ethical use and confidentiality. Requests must be directed to the Corresponding Author and are subject to final approval by the Principal Investigator and the Ethics Committee of Karamanoğlu Mehmetbey University.All shared data will be anonymized and stripped of any identifying information to protect participant privacy.
URL: https://www.kmu.edu.tr